CLINICAL TRIAL: NCT03408353
Title: MERIT (Mammography, Early Detection Biomarkers, Risk Assessment, and Imaging Technologies) Cohort
Brief Title: Mammography, Early Detection Biomarkers, Risk Assessment, and Imaging Technologies, MERIT Study
Status: Recruiting | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: PA17-0584; NCI-2020-07361 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PA17-0584 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2017-12-11; First posted 2018-01-24 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Breast Carcinoma
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational (mammography, questionnaires, blood collection): Participants complete questionnaires over 15-25 minutes about personal and family history of cancer, health status, breast cancer risk factors, diet, weight gain, and physical activity, and undergo collection of blood samples at baseline and then annually for 5 years. Participants also undergo standard of care mammography at baseline and then annually for 5 years.
  Interventions: Procedure: Biospecimen Collection; Procedure: Mammography; Other: Questionnaire Administration

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo collection of blood samples
Procedure: Mammography — Undergo standard of care mammography
Other: Questionnaire Administration — Complete questionnaires

SUMMARY:
This study collects mammogram images, blood samples, and clinical information from women undergoing routine screening mammograms. Creating a bank of blood samples and a database of clinical and risk information may be used in future research related to breast cancer, other cancers, and women's health.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To establish a longitudinal cohort (n=10,000) of women who undergo routine annual mammography screening with follow-up for at least five years for each study participant or until breast cancer diagnosis.

II. To create a repository of blood specimens from the cohort to use for biomarker discovery and validation.

III. To create a comprehensive integrated database of imaging, clinical data, health measurements, and questionnaire data on the study participants.

OUTLINE:

Participants complete questionnaires over 15-25 minutes about personal and family history of cancer, health status, breast cancer risk factors, diet, weight gain, and physical activity, and undergo collection of blood samples at baseline and then annually for 5 years. Participants also undergo standard of care mammography at baseline and then annually for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to participate in the study and ability to provide informed consent
* Willingness to complete a questionnaire and to provide a blood sample at the initial visit and at follow up annual visits
* Undergoing a screening mammogram at participating sites. Subjects undergoing routine annual diagnostic mammograms or CEM as part of a screening study are also eligible.

Exclusion Criteria:

* Current or recent (within the prior 6 months) history of breast feeding
* Personal history of breast cancer (ductal breast carcinoma in situ [DCIS] or invasive breast cancer)
* Personal history of any other cancer (excluding in-situ, stage 0, and non-melanoma skin cancers and other pre-cancerous conditions) treated within the last 5 years.

Ages: 25 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants receiving screening mammograms at MD Anderson site
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2017-09-15 (Actual); Primary Completion 2027-04-30 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Creation of a repository of blood specimens and database of imaging, clinical data, health measurements, and questionnaire data | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Jessica W Leung, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: The University of Texas MD Anderson Cancer Center Official Website — http://www.mdanderson.org